CLINICAL TRIAL: NCT00982020
Title: A Long-Term, Open-Label, Safety Study of Oral Olanzapine in Adolescents With Bipolar I Disorder (Manic or Mixed Episodes) or Schizophrenia
Brief Title: Study in Adolescents With Schizophrenia or Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12117; F1D-MC-HGMX (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-09-15; First posted 2009-09-22 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Bipolar I Disorder; Schizophrenia
Keywords: safety; schizophrenia; bipolar I (manic or mixed); adolescents; weight management
MeSH Terms: conditions — Schizophrenia; Mania | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olanzapine/standard behavioral weight intervention (Experimental)
  Interventions: Drug: Olanzapine; Behavioral: Standard behavioral weight intervention
- Olanzapine/intense behavioral weight intervention (Experimental)
  Interventions: Drug: Olanzapine; Behavioral: Intense behavioral weight intervention

INTERVENTIONS:
Drug: Olanzapine — 2.5 milligrams (mg) to 20 mg given orally, daily for 52 weeks
  Other Names: Zyprexa; LY170053
Behavioral: Standard behavioral weight intervention — One time counseling and basic counseling information on healthy eating and exercise habits at randomization visit only.
  Arms: Olanzapine/standard behavioral weight intervention
Behavioral: Intense behavioral weight intervention — Counseling provided at randomization and at all subsequent study visits by appropriately trained individual regarding healthy lifestyle habits. Participants also provided with simple tools to help enable healthy eating and exercise habits.
  Arms: Olanzapine/intense behavioral weight intervention

SUMMARY:
Open-label safety study of oral olanzapine treatment in adolescents, aged 13 to 17 years, with bipolar I disorder (manic or mixed episodes) or schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of bipolar I disorder and display an acute manic or mixed episode (with or without psychotic features) or a diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM-IV-TR)and confirmed by the Kiddie Schedule for Affective Disorders and Schizophrenia for School Aged Children-Present and Lifetime (K-SADS-PL).
* Participants with a diagnosis of schizophrenia must obtain a Brief Psychiatric Rating Scale for Children (BPRS-C) total score >30, with a minimum score of 3 on at least one of the following items at both screening and randomization - hallucinations, delusions, peculiar fantasies.
* Participants with a diagnosis of bipolar I disorder must have a Young Mania Rating Scale (YMRS) total score greater than or equal to 15 at both screening and randomization.
* Has given assent (when applicable); and has a parent or authorized legal representative who has given informed consent, is reliable, has a level of understanding sufficient to permit participant to perform all tests and examinations required by the protocol, and understands the nature of the study.

Exclusion Criteria:

* History of mental retardation, current comorbid autism, or current comorbid Pervasive Developmental Disorder.
* Have DSM-IV-TR substance (except nicotine and caffeine) dependence within the past 30 days prior to randomization.
* Been judged clinically to be at any suicidal risk.
* History of allergic reaction or hypersensitivity to olanzapine.
* Receiving current pharmaceutical treatment for weight management or are participating in a structured behavioral diet and/or exercise weight loss program.
* Other antipsychotics, mood stabilizers, or anticonvulsants (for mood stabilization) used for the primary study conditions (bipolar I disorder or schizophrenia)
* Have acute, serious, or unstable medical conditions
* Have any illness such that death is anticipated within 1 year or intensive care unit hospitalization for the illness is anticipated within 12 months (365 days).
* Have had one or more seizures without a clear and resolved etiology.
* Baseline alanine aminotransferase (ALT) values greater than or equal to 2 times the upper limit of normal (ULN) of the performing laboratory or aspartate aminotransferase (AST) values greater than or equal to 2 times the ULN or total bilirubin values greater than or equal to 1.5 times the ULN at screening.
* Have leukopenia or history of leukopenia without a clear and resolved etiology or known history of agranulocytosis (absolute neutrophil count <500 cubic millimeter [mm^3], <0.5 GI/L, or <0.5 10E^3/microliters [μL]) during the participant's lifetime.
* Prolactin level of >200 nanograms per milliliter (ng/mL) [>200 micrograms per liter (ug/L), or >4228 milli-International unit per liter (mIU/L)] at screening.
* Have QTc (Bazett's) >450 milliseconds (males) or >460 milliseconds (females) at screening.
* Previously been randomized in this study and/or participated in a clinical trial of another investigational drug, including olanzapine, within 1 month (30 days) prior to screening.
* Currently prescribed olanzapine for greater than or equal to 5 days within 1 month (30 days) prior to screening.
* Are investigator site personnel directly affiliated with this study and/or their immediate families OR are employed by or representatives of Lilly.
* Pregnant or nursing.
* Have received treatment within the last 30 days with an investigational new drug that has not received regulatory approval for any indication at the time of study entry.
* Treatment with clozapine within 14 days prior to randomization.
* Participants who have used olanzapine (that is, oral olanzapine, intramuscular [IM] olanzapine, or olanzapine orally disintegrating tablets) and have had treatment withdrawn due to clinically significant and/or intolerable adverse effects, or who have exhibited a lack of efficacy/response to treatment to olanzapine including treatment resistance.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 203 (Actual)
Dates: Start 2009-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lauderhill, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloomfield Hills, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
- Poland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caguas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- Russia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lipetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petrozavodsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saratov

REFERENCES:
- [Derived] Detke HC, DelBello MP, Landry J, Hoffmann VP, Heinloth A, Dittmann RW. A 52-Week Study of Olanzapine with a Randomized Behavioral Weight Counseling Intervention in Adolescents with Schizophrenia or Bipolar I Disorder. J Child Adolesc Psychopharmacol. 2016 Dec;26(10):922-934. doi: 10.1089/cap.2016.0010. Epub 2016 Sep 27. PMID 27676420

RESULTS

PARTICIPANT FLOW:
Groups:
- Olanzapine/Standard Behavioral Weight Intervention: Olanzapine: 2.5 milligrams (mg) to 20 mg given orally, daily for 52 weeks. Standard behavioral weight intervention: One time counseling and basic counseling information on healthy eating and exercise habits at randomization visit only
- Olanzapine/Intense Behavioral Weight Intervention: Olanzapine: 2.5 mg to 20 mg given orally, daily for 52 weeks. Intense behavioral weight intervention: Counseling provided at randomization and at all subsequent study visits by appropriately trained individual regarding healthy lifestyle habits. Participants also provided with simple tools to help enable healthy eating and exercise habits
Period: Overall Study
Arm/Group | Olanzapine/Standard Behavioral Weight Intervention | Olanzapine/Intense Behavioral Weight Intervention
Started | 102 | 101
Received at Least 1 Dose of Study Drug | 102 | 101
Completed | 45 | 37
Not Completed | 57 | 64
Not completed — Adverse Event | 19 | 15
Not completed — Withdrawal by Subject | 11 | 14
Not completed — Lost to Follow-up | 5 | 11
Not completed — Lack of Efficacy | 10 | 4
Not completed — Parent/Caregiver Decision | 5 | 5
Not completed — Treatment Non-compliance | 3 | 6
Not completed — Physician Decision | 2 | 5
Not completed — Entry Criteria Not Met | 2 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Clinical Relapse | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug
Groups:
- Olanzapine/Standard Behavioral Weight Intervention: Olanzapine: 2.5 mg to 20 mg given orally, daily for 52 weeks.
  Standard behavioral weight intervention: One time counseling and basic counseling information on healthy eating and exercise habits at randomization visit only
- Total: Total of all reporting groups
Arm/Group | Olanzapine/Standard Behavioral Weight Intervention | Olanzapine/Intense Behavioral Weight Intervention | Total
Number analyzed (Participants) | 102 | 101 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.86 (1.49) | 15.66 (1.52) | 15.76 (1.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 47 | 97
  Male | 52 | 54 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 9 | 24
  Not Hispanic or Latino | 87 | 92 | 179
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 14 | 26
  White | 84 | 80 | 164
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 2 | 1 | 3
  Poland | 6 | 12 | 18
  Russian Federation | 28 | 27 | 55
  United States | 53 | 54 | 107
  Puerto Rico | 13 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to 52 Weeks in Body Mass Index (BMI) for All Participants
Time Frame: Baseline, 52 weeks
Population: All randomized participants who received at least one dose of study drug. Mixed model repeated measures (MMRM) methodology used.
Measure: Least Squares Mean (Standard Error); unit: kilograms per meter squared (kg/m^2)
Arm/Group | Olanzapine/Standard Behavioral Weight Intervention | Olanzapine/Intense Behavioral Weight Intervention
Number analyzed (Participants) | 102 | 101
kilograms per meter squared (kg/m^2) | 3.64 (.39) | 2.83 (.40)
Statistical Analysis 1: Comparison: Olanzapine/Standard Behavioral Weight Intervention vs Olanzapine/Intense Behavioral Weight Intervention; Test type: Superiority or Other; p = 0.150, Mixed Models Analysis — The threshold for statistical significance was 0.05; Mixed model repeated measures analysis terms included baseline BMI, baseline age, gender, intervention group, visit, region, intervention group*visit

2. Secondary Outcome: Mean Change From Baseline to Endpoint in Body Mass Index (BMI) for Participants With Duration of Treatment of at Least 6 Months
Time Frame: Baseline, 52 weeks
Population: All randomized participants who received at least one dose of study drug and who had at least 6 months of data. Last observation carried forward (LOCF) methodology.
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Olanzapine/Standard Behavioral Weight Intervention | Olanzapine/Intense Behavioral Weight Intervention
Number analyzed (Participants) | 54 | 55
kg/m^2 | 3.36 (0.41) | 2.99 (0.40)
Statistical Analysis 1: Comparison: Olanzapine/Standard Behavioral Weight Intervention vs Olanzapine/Intense Behavioral Weight Intervention; Test type: Superiority or Other; p = 0.520, ANCOVA — The threshold for statistical significance was 0.05; ANCOVA model terms included: baseline, baseline age, gender, intervention group, and region

3. Secondary Outcome: Time to Event for 7%, 15%, and 25% Weight Gain for All Participants
Description: Kaplan-Meier methodology used to estimate time to event. Participants who never reached the target weight gain contributed to the set of patients at risk up to the point at which they discontinued from the study and were then censored (i.e., removed from the risk set).
Time Frame: Baseline up to 52 weeks
Population: 65 participants (32%; 34% in Standard Group [SG], 30% in Intense Group [IG]) did not meet 7% weight gain criterion [WGC] by the time they discontinued.
  122 participants (60%; 58% in SG, 62% in IG) did not meet 15% WGC by the time they discontinued.
  161 participants (79%; 76% in SG, 82% in IG) did not meet 25% WGC by the time they discontinued.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Olanzapine/Standard Behavioral Weight Intervention | Olanzapine/Intense Behavioral Weight Intervention
Number analyzed (Participants) | 102 | 101
days
  Time to First 7% Weight Gain | 57 [44.00 to 84.00] | 57 [44.00 to 84.00]
  Time to First 15% Weight Gain | 197 [140.00 to 359.00] | 198 [141.00 to NA] — There was an insufficient number of events of 15% weight gain in the Intense group to compute this statistic.
  Time to First 25% Weight Gain | NA [NA to NA] — There was an insufficient number of events of 25% weight gain in the Standard group to compute these statistics. | NA [NA to NA] — There was an insufficient number of events of 25% weight gain in the Intense group to compute these statistics.

4. Secondary Outcome: Mean Change From Baseline to 52 Weeks in Adolescent Structured Young Mania Rating Scale (YMRS) for Participants With Bipolar I Disorder
Description: The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 (symptom not present) to 60 (symptom extremely severe).
Time Frame: Baseline, 52 weeks
Population: All randomized participants with bipolar I disorder, who received at least one dose of study drug. Mixed model repeated measures (MMRM) methodology.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Olanzapine/Standard Behavioral Weight Intervention | Olanzapine/Intense Behavioral Weight Intervention
Number analyzed (Participants) | 58 | 58
units on a scale | -17.66 (1.75) | -12.05 (1.92)
Statistical Analysis 1: Comparison: Olanzapine/Standard Behavioral Weight Intervention vs Olanzapine/Intense Behavioral Weight Intervention; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis — Threshold for statistical significance was 0.05; MMRM analysis terms included baseline, intervention group, visit, region, and intervention group*visit

5. Secondary Outcome: Mean Clinical Global Impression of Improvement (CGI-I) at 52 Weeks for All Participants
Description: The Clinical Global Impression of Improvement (CGI-I) is used by the clinician to record the improvement of illness at the time of assessment. The score ranges from 1 (very much improved) to 7 (very much worse).
Time Frame: 52 weeks
Population: All randomized participants who received at least one dose of study drug. Mixed model repeated measures (MMRM) methodology.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Olanzapine/Standard Behavioral Weight Intervention | Olanzapine/Intense Behavioral Weight Intervention
Number analyzed (Participants) | 102 | 101
units on a scale | 2.04 (0.15) | 2.29 (0.16)
Statistical Analysis 1: Comparison: Olanzapine/Standard Behavioral Weight Intervention vs Olanzapine/Intense Behavioral Weight Intervention; Test type: Superiority or Other; p = 0.266, Mixed Models Analysis — The threshold for statistical significance was 0.05; MMRM analysis terms included intervention group, visit, region, and intervention group*visit

6. Secondary Outcome: Mean Change From Baseline to 52 Weeks in Waist Circumference for All Participants
Time Frame: Baseline, 52 weeks
Population: All randomized participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: centimeters (cm)
Arm/Group | Olanzapine/Standard Behavioral Weight Intervention | Olanzapine/Intense Behavioral Weight Intervention
Number analyzed (Participants) | 102 | 101
centimeters (cm) | 7.22 (1.06) | 7.31 (1.11)
Statistical Analysis 1: Comparison: Olanzapine/Standard Behavioral Weight Intervention vs Olanzapine/Intense Behavioral Weight Intervention; Test type: Superiority or Other; p = 0.954, Mixed Models Analysis — The threshold for statistical significance was 0.05; MMRM analysis terms included baseline, baseline age, gender, intervention group, visit, region, and intervention group*visit

7. Secondary Outcome: Mean Change From Baseline to 52 Weeks in Clinical Global Impression - Severity (CGI-S) for All Participants
Description: The CGI-S is used by the clinician to record the severity of illness at the time of assessment. The score ranges from 1 = normal, not at all ill to 7 = among the most extremely ill.
Time Frame: Baseline, 52 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Olanzapine/Standard Behavioral Weight Intervention | Olanzapine/Intense Behavioral Weight Intervention
Number analyzed (Participants) | 102 | 101
units on a scale | -2.06 (0.14) | -1.74 (0.14)
Statistical Analysis 1: Comparison: Olanzapine/Standard Behavioral Weight Intervention vs Olanzapine/Intense Behavioral Weight Intervention; Test type: Superiority or Other; p = 0.103, Mixed Models Analysis — Threshold for statistical significance was 0.05; MMRM analysis terms included baseline, intervention group, visit, region, and intervention group*visit

8. Secondary Outcome: Mean Change From Baseline to 52 Weeks in Anchored Version of the Brief Psychiatric Rating Scale for Children (BPRS-C) for Participants With Schizophrenia
Description: The BPRS-C characterizes psychopathology. A total of 21 items are rated on a scale from 0 (not present) to 6 (extremely severe) with a total score ranging from 0 to 126. A decrease in score indicates a reduction in psychopathology.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with schizophrenia who received at least one dose of study drug. Mixed model repeated measures (MMRM) methodology.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Olanzapine/Standard Behavioral Weight Intervention: Olanzapine: 2.5 mg to 20 mg given orally, daily for 52 weeks Standard behavioral weight intervention: One time counseling and basic counseling information on healthy eating and exercise habits at randomization visit only
- Olanzapine/Intense Behavioral Weight Intervention: Olanzapine: 2.5 mg to 20 mg given orally, daily for 52 weeks Intense behavioral weight intervention: Counseling provided at randomization and at all subsequent study visits by appropriately trained individual regarding healthy lifestyle habits. Participants also provided with simple tools to help enable healthy eating and exercise habits
Arm/Group | Olanzapine/Standard Behavioral Weight Intervention | Olanzapine/Intense Behavioral Weight Intervention
Number analyzed (Participants) | 44 | 43
units on a scale | -28.00 (2.83) | -30.96 (2.67)
Statistical Analysis 1: Comparison: Olanzapine/Standard Behavioral Weight Intervention vs Olanzapine/Intense Behavioral Weight Intervention; Test type: Superiority or Other; p = 0.436, Mixed Models Analysis — The threshold for statistical significance was 0.05; MMRM analysis terms included baseline, intervention group, visit, region, and intervention group*visit

ADVERSE EVENTS:
Groups:
- Olanzapine/Standard Behavioral Weight Intervention: Olanzapine: 2.5mg to 20mg given orally, daily for 52 weeks
  Standard behavioral weight intervention: One time counseling and basic counseling information on healthy eating and exercise habits at randomization visit only
- Olanzapine/Intense Behavioral Weight Intervention: Olanzapine: 2.5mg to 20mg given orally, daily for 52 weeks
  Intense behavioral weight intervention: Counseling provided at randomization and at all subsequent study visits by appropriately trained individual regarding healthy lifestyle habits. Participants also provided with simple tools to help enable healthy eating and exercise habits.
Arm/Group | Olanzapine/Standard Behavioral Weight Intervention | Olanzapine/Intense Behavioral Weight Intervention
Serious Adverse Events (participants affected / at risk) | 13/102 | 20/101
Other Adverse Events (participants affected / at risk) | 81/102 | 81/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine/Standard Behavioral Weight Intervention (N=102) | Olanzapine/Intense Behavioral Weight Intervention (N=101)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 1 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neuroleptic malignant syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (2)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Bipolar i disorder (Psychiatric disorders) | 0 (0) | 4 (4)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 4 (5)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Schizophrenia, paranoid type (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 3 (3) | 2 (2)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Olanzapine/Standard Behavioral Weight Intervention (N=102) | Olanzapine/Intense Behavioral Weight Intervention (N=101)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 4 (4)
Vomiting (Gastrointestinal disorders) | 7 (8) | 4 (7)
Fatigue (General disorders) | 9 (10) | 6 (6)
Nasopharyngitis (Infections and infestations) | 14 (16) | 11 (11)
Blood creatine phosphokinase increased (Investigations) | 7 (9) | 5 (6)
Blood insulin increased (Investigations) | 10 (11) | 7 (7)
Weight increased (Investigations) | 31 (31) | 21 (21)
Increased appetite (Metabolism and nutrition disorders) | 16 (16) | 13 (14)
Dizziness (Nervous system disorders) | 7 (7) | 2 (2)
Headache (Nervous system disorders) | 19 (49) | 20 (30)
Sedation (Nervous system disorders) | 8 (8) | 3 (5)
Somnolence (Nervous system disorders) | 19 (22) | 24 (28)
Anxiety (Psychiatric disorders) | 6 (6) | 3 (4)
Dysmenorrhoea (Reproductive system and breast disorders) | 3/50 (18) | 1/47 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days